CLINICAL TRIAL: NCT05657093
Title: "Effects of Beetroot Juice os Sport Performane in Elite Swimmers. A Randomized Clinical Trial"
Brief Title: Effect of the Beetroot Juice in Portuguese Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Universidad Politecnica de Madrid (Other); Instituto Politécnico de Bragança (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 79/2022
Record Dates: First submitted 2022-12-01; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Ergogenics
Keywords: swimming; beet; swim; nitrate; intermittent sports; ergogenic aids

STUDY DESIGN:
Intervention Model Description: Parallel allocation was carried out in the two groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blinded (Participant, Investigator and Outcomes Assessor) The participant was blinded not knowing the treatment to which he was submitted, investigator and outcome assessor responsible for collecting the results, without commenting on the group from which the subject came.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Active Comparator): The swimmers ingested a shot of Beet-It 70 ml beetroot juice (BJ)) 3 hours before undergoing a 2x6x100m crawl intermittent maximal speed performance test.
  Interventions: Dietary Supplement: Beetroot Juice; Combination Product: Placebo
- Placebo (Placebo Comparator): The swimmers ingested a shot of Beet-It (70 ml placebo (PL)) 3 hours before undergoing a 2x6x100m crawl intermittent maximal speed performance test.
  Interventions: Dietary Supplement: Beetroot Juice; Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — The swimmers drank 3 hours before the test, mL70 of BJ (containing mmol6.4 of NO-3) (Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) or PLA (0.04 mmol of NO-3)
Combination Product: Placebo — The swimmers drank 3 hours before the test, mL70 of BJ (containing mmol6.4 of NO-3) (Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) or PLA (0.04 mmol of NO-3)

SUMMARY:
Objective: To investigate whether an acute intake of beet juice (BJ) improved the factors of total and split times (performance), stroke frequency and CMJ (biomechanics), lactate and HR (physiology) and RPE-TQR (psychophysiological) in a repeated (performance), stroke frequency and CMJ (biomechanics), lactate and HR (physiology) and RPE-TQR (psychophysiological) in a repeated maximal speed swimming effort in elite swimmers.

Methods: A total of 18 elite swimmers participated in this randomized, double-blind study. In 2 different trials, swimmers ingested a Beet-It injection (70 ml placebo (PL) or a Beet-It injection of 70 ml beet juice (BJ)) 3 hours before undergoing a 2x6x100 m intermittent maximal speed crawl performance test.

ELIGIBILITY:
Inclusion Criteria:

1. - national and international level swimmers
2. - healthy swimmers
3. - no breakfast
4. - 48 hours with restricted diet of: other sports supplements and beetroot-rich foods

Exclusion Criteria:

1. -be on medication
2. - having had breakfast
3. - have brushed your teeth

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-05-07 (Actual)

PRIMARY OUTCOMES:
Lactate concentration | 3 hours post-dose of Beetroot juice or Placebo
  After qeach even series of 100m (2nd, 4th, 6th and 3' rest), their finger was wiped dry and their blood lactate concentration was measured with a Lactate Pro2 portable analyzer 1 minute after completing each 100m series.
Rate of Perceived Exertion | 3 hours after ingestion of the beetroot juice
  During every 100m, they were asked how much effort they had exerted using the subjective RPE scale as in other studies with BJ and swimming.
Recovery Total Quality Scale | 3 hours after ingestion of the beetroot juice
  Before the swimmers performed the next 100m, they were asked how recovered they felt, using another subjective TQR scale.
Total Time | 3 hours after ingestion of the beetroot juice
  The complete 2x6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the total times, with the program KINOVEA 0.9.5.
Parcial Time | 3 hours after ingestion of the beetroot juice
  The complete 2x6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the split times, with the KINOVEA 0.9.5 program.
Counter Movement Jump | 3 hours after ingestion of the beetroot juice
  Swimmers completed three repetitions of CMJ with hands on waist using an infrared jumping system (Optojump Next, Microgate, Bolzano, Italy)

SECONDARY OUTCOMES:
Stroke rate | from the day of randomization to the last day of the intervention: up to day 7
  The complete 2x6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the stroke rate, with the KINOVEA 0.9.5 program.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Madrid, Pozuelo de Alarcón, Spain

REFERENCES:
- [Result] Moreno B, Veiga S, Sanchez-Oliver AJ, Dominguez R, Morencos E. Analysis of Sport Supplement Consumption by Competitive Swimmers According to Sex and Competitive Level. Nutrients. 2022 Aug 6;14(15):3218. doi: 10.3390/nu14153218. PMID 35956394
- [Result] Senefeld JW, Wiggins CC, Regimbal RJ, Dominelli PB, Baker SE, Joyner MJ. Ergogenic Effect of Nitrate Supplementation: A Systematic Review and Meta-analysis. Med Sci Sports Exerc. 2020 Oct;52(10):2250-2261. doi: 10.1249/MSS.0000000000002363. PMID 32936597
- [Result] Zamani H, de Joode MEJR, Hossein IJ, Henckens NFT, Guggeis MA, Berends JE, de Kok TMCM, van Breda SGJ. The benefits and risks of beetroot juice consumption: a systematic review. Crit Rev Food Sci Nutr. 2021;61(5):788-804. doi: 10.1080/10408398.2020.1746629. Epub 2020 Apr 15. PMID 32292042
- [Result] Berjisian E, McGawley K, Saunders B, Dominguez R, Koozehchian MS, de Oliveira CVC, Rafiei R, Miraftabi H, Sarshin A, Naderi A. Acute effects of beetroot juice and caffeine co-ingestion during a team-sport-specific intermittent exercise test in semi-professional soccer players: a randomized, double-blind, placebo-controlled study. BMC Sports Sci Med Rehabil. 2022 Mar 29;14(1):52. doi: 10.1186/s13102-022-00441-1. PMID 35351196
- [Result] Jonvik KL, Hoogervorst D, Peelen HB, de Niet M, Verdijk LB, van Loon LJC, van Dijk JW. The impact of beetroot juice supplementation on muscular endurance, maximal strength and countermovement jump performance. Eur J Sport Sci. 2021 Jun;21(6):871-878. doi: 10.1080/17461391.2020.1788649. Epub 2020 Jul 21. PMID 32594854
- [Result] Morais JE, Silva AJ, Garrido ND, Marinho DA, Barbosa TM. The transfer of strength and power into the stroke biomechanics of young swimmers over a 34-week period. Eur J Sport Sci. 2018 Jul;18(6):787-795. doi: 10.1080/17461391.2018.1453869. Epub 2018 Mar 24. PMID 29577827
- [Result] Esen O, Dominguez R, Karayigit R. Acute Beetroot Juice Supplementation Enhances Intermittent Running Performance but Does Not Reduce Oxygen Cost of Exercise among Recreational Adults. Nutrients. 2022 Jul 11;14(14):2839. doi: 10.3390/nu14142839. PMID 35889796